CLINICAL TRIAL: NCT01898273
Title: Phase 2, Open-Label, Imaging Trial of I-124-CLR1404 in Patients With Newly Diagnosed or Recurrent Glioblastoma
Brief Title: Imaging Trial With I-124-CLR1404 in Patients With Newly Diagnosed or Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DCL-13-002
Record Dates: First submitted 2013-07-08; First posted 2013-07-12 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Glioblastoma
Keywords: Glioma; Glioblastoma Multiforme; PET; Imaging; Radiopharmaceutical; Diagnostic
MeSH Terms: conditions — Glioblastoma; Glioma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): I-124-CLR1404, open-label
  Interventions: Drug: I-124-CLR1404

INTERVENTIONS:
Drug: I-124-CLR1404 — single-dose, intravenous
  Other Names: I-124-NM404

SUMMARY:
The primary objective of this trial is to determine the optimal dose and imaging time point(s) of I-124-CLR1404 in subjects with newly diagnosed and recurrent glioma to be used in future trials.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed glioblastoma or recurrent/suspected recurrent glioblastoma
* scheduled to undergo a clinically-indicated surgery or biopsy (specific cohorts)
* ECOG performance status of 0 to 2 (Appendix C)
* 18 years of age or older
* has the initiative and means to be compliant with the protocol and be within geographical proximity to make the required study visits
* has the ability to read, understand and provide written informed consent for the initiation of any study related procedures (or legal representative)
* if female of childbearing potential must have a negative pregnancy test within 24 hours of enrollment
* Women of childbearing potential and men who are able to father a child, must agree to use an effective method of contraception (e.g., oral contraceptives, double-barrier methods such as a condom and a diaphragm, intrauterine device, Norplant, Depo-Provera) during the study and for 45 days following the last dose of the study drug.

Exclusion Criteria:

* ongoing grade 2 or greater toxicities due to previous therapies. However, tolerable grade 2 adverse (e.g. neuropathy) events may be allowed at the discretion of the investigator.
* has following laboratory abnormalities

  * Platelets < 100,000/μL
  * WBC < 3000/μL
  * Hematocrit < 22%
  * Serum creatinine > 2.5 mg/dL
  * ALT > 1.5 x ULN
  * Bilirubin > 1.5 x ULN
* ongoing chronic immunosuppressive therapy
* history of hypersensitivity to iodine
* any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise subject safety or interfere with the evaluation of the safety of the test drug
* women of childbearing potential, or men who are able to father a child, unwilling to use a medically acceptable method of contraception during the trial
* pregnancy or breast-feeding
* inability to comply with the protocol
* use of any investigational drug within 4 weeks of dosing (unless a longer time period is required by local regulations or the investigational agent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Optimal Imaging Parameters - Dose | 8 days
  Up to two dose levels (5 mCi and 7.5 mCi) will be evaluated in conjunction with multiple imaging time points to determine the optimal parameters for PET/CT brain imaging. Dosing will begin at 5 mCi and if the images are deemed inadequate, as assessed by count statistics and image quality, the 7.5 mCi dose level will be evaluated.

SECONDARY OUTCOMES:
Optimal Imaging Parameters - Imaging Time Point | 8 days
  Multiple imaging time points (Day 2, Day 3, and Day 4-8) will be evaluated to determine the optimal parameters for PET/CT brain imaging.

CONTACTS AND LOCATIONS:
Overall Officials: John Kuo, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Jana Portnow, MD, Principal Investigator — City of Hope Medical Center; Abass Alavi, MD, Principal Investigator — University of Pennsylvania
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin